CLINICAL TRIAL: NCT00033163
Title: A Randomized, Phase II, Controlled Trial Comparing the Efficacy of Adefovir Dipivoxil and Tenofovir Disoproxil Fumarate for the Treatment of Lamivudine-Resistant Hepatitis B Virus in Subjects Who Are Co-Infected With HIV
Brief Title: A Comparison of Adefovir and Tenofovir for the Treatment of Lamivudine-Resistant Hepatitis B Virus in People With HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: A5127; 10678 (Registry Identifier: DAIDS ES); ACTG A5127; AACTG A5127
Record Dates: First submitted 2002-04-08; First posted 2002-04-09 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Hepatitis B
Keywords: Antiviral Agents; Hepatitis B; Drug Resistance, Microbial; Lamivudine; DNA, Viral; Hepatitis B Virus; Adefovir dipivoxil; Tenofovir disoproxil fumarate; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Hepatitis B | interventions — adefovir dipivoxil; Tenofovir

INTERVENTIONS:
Drug: Adefovir dipivoxil
Drug: Tenofovir disoproxil fumarate

SUMMARY:
Control of hepatitis B virus (HBV) infection can be difficult in HIV infected people who have taken the antiviral lamivudine (3TC). These people may have HBV that has become resistant to 3TC. Adefovir dipivoxil (ADV) has shown promising anti-HBV activity in clinical trials; tenofovir disoproxil fumarate (TDF) is used to treat HIV and may also be effective against HBV. The purpose of this study is to find out if adding ADV or TDF to a highly active antiretroviral therapy (HAART) regimen that includes 3TC has an effect on HBV infection in patients coinfected with HIV and HBV. The tolerability and safety of these drugs will be examined.

DETAILED DESCRIPTION:
HBV presents a worldwide health crisis and is difficult to treat when a patient's HBV strain is no longer responsive to 3TC. Given the significant incidence of 3TC-resistant HBV in patients receiving this drug as part of an antiretroviral regimen, other agents with anti-HBV activity are needed. ADV has shown promising anti-HBV activity in preclinical assessments and in Phase I, II, and III clinical trials. TDF, developed for the treatment of HIV infection, has in vitro activity against HBV. This study will compare TDF/3TC combination therapy with ADV/3TC combination therapy to determine which treatment regimen is more effective in patients coinfected with HBV and HIV.

This study will include two populations of patients. Patients in Population A are on stable HAART that includes TDF and will either be in Group I (compensated liver disease) or Group II (decompensated liver disease). All patients in Population A will be randomly assigned to one of two arms: Arm 1 patients will receive 10 mg ADV daily and TDF placebo; Arm 2 patients will receive ADV placebo and 300 mg TDF. Patients in Population B are on stable HAART and have never taken TDF as part of their HAART. Population B patients will receive 300 mg TDF daily during the course of the study.

Study visits will occur every 4 weeks for the 96-week study period. Targeted clinical and medication assessments and blood work assessing clotting time, liver function, and blood chemistry will be conducted at each study visit. HIV and HBV DNA viral load will be tested every 12 weeks. CD4 cell counts will be tested at Weeks 24, 48, 72, and 96.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* HIV infected
* HBV infected
* Serum HBV DNA of 100,000 copies/ml or greater
* Positive for serum hepatitis B surface antigen (HBsAg) within 12 weeks prior to study entry
* Agree to use acceptable methods of contraception
* Serum alpha-fetoprotein (AFP) of 50 ng/ml or less within 30 days of study entry. If AFP is greater than 50 ng/ml, the patient must have an imaging study of the liver showing no tumor within 30 days prior to study entry

Inclusion Criteria for Population A:

* Uninterrupted stable HAART regimen at study entry for at least 12 continuous weeks prior to study entry
* HIV viral load of 10,000 copies/ml or less within 12 weeks of study entry

Inclusion Criteria for Population A, Group I:

* Compensated liver disease
* Child-Pugh-Turcotte (CPT) score of less than 7

Exclusion Criteria for Population A, Group I:

* Excess fluid in the space between the membranes lining the abdomen and abdominal organs (ascites)
* Gastrointestinal (variceal) bleeding
* Brain and nervous system damage as a result of liver disease
* Abnormal blood clotting time

Inclusion Criteria for Population A, Group II:

* Decompensated liver disease
* CPT score of 7-12

Inclusion Criteria for Population B:

* Prior HAART regimen
* Never taken TDF as part of HAART regimen
* Serum HBV DNA of 100,000 copies/ml or greater within 12 weeks of study entry
* HIV viral load of greater than 10,000 copies/ml within 12 weeks of study entry
* CPT score less than 13

Exclusion Criteria

* Serious kidney problems within the last 12 months
* Allergic or sensitive to ADV or TDF
* Active hepatitis C virus (HCV) disease or unknown HCV status within 24 weeks of study entry
* Any medical or mental illness that, in the opinion of the investigator, would interfere with the protocol
* Past or current alcohol or drug abuse that would affect the protocol
* Malignancy that, in the opinion of the investigator, would make the patient unsuitable for the study
* Certain anti-HBV drugs within 90 days of study entry or expected use of these agents during the course of the study
* Drugs that may damage the kidneys within 8 weeks prior to study screening or expected use of these agents during the course of the study
* Systemic corticosteroids within 90 days of study entry
* Current use of drugs containing pivalic acid
* Certain investigational anti-HIV agents
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Polsky, MD, Study Chair — St. Luke's-Roosevelt Hospital Center; Marion Peters, MD, Study Chair — University of California, San Francisco
Locations (15):
- United States (15):
  - UC Davis Medical Center, Sacramento, California
  - Univ. of California Davis Med. Ctr., ACTU, Sacramento, California
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell CRS, New York, New York
  - Weill Med. College of Cornell Univ., The Cornell CTU, New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Benhamou Y, Bochet M, Thibault V, Di Martino V, Caumes E, Bricaire F, Opolon P, Katlama C, Poynard T. Long-term incidence of hepatitis B virus resistance to lamivudine in human immunodeficiency virus-infected patients. Hepatology. 1999 Nov;30(5):1302-6. doi: 10.1002/hep.510300525. PMID 10534354
- [Background] Benhamou Y, Bochet M, Thibault V, Calvez V, Fievet MH, Vig P, Gibbs CS, Brosgart C, Fry J, Namini H, Katlama C, Poynard T. Safety and efficacy of adefovir dipivoxil in patients co-infected with HIV-1 and lamivudine-resistant hepatitis B virus: an open-label pilot study. Lancet. 2001 Sep 1;358(9283):718-23. doi: 10.1016/s0140-6736(01)05840-8. PMID 11551579
- [Background] Dieterich DT. HIV and hepatitis B virus: options for managing coinfection. Top HIV Med. 2003 Jan-Feb;11(1):16-9. PMID 12717046
- [Background] Rockstroh JK. Management of hepatitis B and C in HIV co-infected patients. J Acquir Immune Defic Syndr. 2003 Sep;34 Suppl 1:S59-65. doi: 10.1097/00126334-200309011-00009. PMID 14562859
- [Background] Thio CL. Hepatitis B in the human immunodeficiency virus-infected patient: epidemiology, natural history, and treatment. Semin Liver Dis. 2003 May;23(2):125-36. doi: 10.1055/s-2003-39951. PMID 12800066
- [Result] Peters MG, Andersen J, Lynch P, Liu T, Alston-Smith B, Brosgart CL, Jacobson JM, Johnson VA, Pollard RB, Rooney JF, Sherman KE, Swindells S, Polsky B; ACTG Protocol A5127 Team. Randomized controlled study of tenofovir and adefovir in chronic hepatitis B virus and HIV infection: ACTG A5127. Hepatology. 2006 Nov;44(5):1110-6. doi: 10.1002/hep.21388. PMID 17058225
- [Derived] Johnson VA, Cramer YS, Rosenkranz SL, Becker S, Klingman KL, Kallungal B, Coakley E, Acosta EP, Calandra G, Saag MS; NIH/NIAID AIDS Clinical Trials Group A5210 Protocol Team. Antiretroviral Activity of AMD11070 (An Orally Administered CXCR4 Entry Inhibitor): Results of NIH/NIAID AIDS Clinical Trials Group Protocol A5210. AIDS Res Hum Retroviruses. 2019 Aug;35(8):691-697. doi: 10.1089/AID.2018.0256. Epub 2019 Jun 18. PMID 31099252